CLINICAL TRIAL: NCT02947906
Title: Investigating the Plantar Pressure Distribution in Patient With Multiple Sclerosis
Brief Title: Plantar Pressure Distribution in Patient With Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, hhotaman, PhD, PT, Hacettepe University
Other Study IDs: G0 16/344
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Gait; Loading; Multiple Sclerosis; Plantar Pressure
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Study group: Participants with multiple sclerosis who able to walk at least 30 meters independently.
  Interventions: Other: No intervention
- Control Group: Healthy participants
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Fifty patients who were referred to receive physiotherapy and 20 healthy volunteers will be participants of the study.Participants with multiple sclerosis will evaluate with the following assessment tools: Modified Ashworth scale will use to evaluation of severity of plantar flexor spasticity. Plantar pressure distribution parameters will assess with dynamic pedobarography.

DETAILED DESCRIPTION:
Fifty patients who were referred to receive physiotherapy at the neurology department of Physiotherapy and Rehabilitation of the Faculty of Health Sciences of Hacettepe University, Ankara with multiple sclerosis and twenty voluntary healthy age matched participants will be the subjects of this study.

Assessment tools described as following: Modified Ashworth scale will use to evaluate of severity of plantar flexor spasticity. Static and dynamic loading parameters will be evaluate with pedobarography.Maximum loading pressure -N/cm2, maximum loading time- ms for; 1st. and 5th metatarsal head, medial and lateral heel and midfoot will be recorded both while the patients standing and walking.

ELIGIBILITY:
Inclusion Criteria:

* Want to participate Individuals with multiple sclerosis who can walk alone for 30 meters Healthy participants who diagnosed no disorders or orthopedic problems.

Exclusion Criteria:

* Want to participate Individuals with multiple sclerosis who can walk alone for 50 meters Healthy participants who diagnosed no disorders or orthopedic problems.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants with multiple sclerosis
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Pedobarography for assessment of foot pressure while standing and walking | Initially evaluation at first minute, Change from initial evaluation to 20th minutes, Change from initial evaluation to 24 hours, Change from initial evaluation to 24 hours and 20 minutes
  Participant stands and walks on system name is pedobarography which records foot pressure. Foot pressure means, gravitational force reflecting from ground at every foot step phase. Newton/cm2 is the unit of measure.

IPD SHARING:
Plan to Share IPD: Undecided